CLINICAL TRIAL: NCT05116735
Title: Biliary Fistula and Late Recurrence of Liver Hydatid Cyst: Role of Cysto-biliary Communication - A Prospective Multicenter Study.
Brief Title: Biliary Fistula and Late Recurrence of Liver Hydatid Cyst: Role of Cysto-biliary Communication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, assistant professour of general and laparoscopic surgery, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hydatid cyst in liver
Record Dates: First submitted 2021-10-29; First posted 2021-11-11 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Liver Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laparoscopic partial cystectomy with omentoplasty (Experimental): laparoscopic partial cystectomy with omentoplasty
  Interventions: Procedure: laparoscopic partial cystectomy with omentoplasty

INTERVENTIONS:
Procedure: laparoscopic partial cystectomy with omentoplasty — laparoscopic partial cystectomy with omentoplasty

SUMMARY:
Purpose : The primary goals of this study were to determine the prevalence and risk factors of occult CBC and recurrence, as well as the relationship between occult cysto-biliary communications manifested as postoperative biliary leakage and recurrence. The secondary goal was to use chemical analysis of hydatid cyst fluid to assess excessive bilirubin and alkaline phosphatase levels as predictors of fistula and recurrence.

Methods: This prospective multi-center experimental and follow-up study of six years duration was conducted at the hepato-biliary pancreatic units of our universities hospitals from September 2010 to September 2016. Initially, 292 patients were included, but only 244 patients enrolled in the final study.

DETAILED DESCRIPTION:
Hydatid cyst disease (HCD) is a zoonotic illness caused by Echinococcus Granulosus that infects humans via ingestion of eggs and primarily affects the liver (50-70%), followed by the lungs, brain, and other viscera . To facilitate consistent diagnosis, treatment, and follow-up, the World Health Organization Informal Working Group on Echinococcosis (WHO-IWGE) arranged a standardized ultrasonography staging based on the cyst's active-transitional-inactive stage .

Various therapy options for hydatid cyst management range from medical treatment alone, which has been shown to be ineffective in curing the condition , to surgical treatment, which is considered the primary therapeutic option [6]. For hydatid cysts, laparoscopic surgery is both safe and successful. Laparoscopic procedures range from conservative procedures such as laparoscopic partial cystectomy and omentoplasty to obliterate the residual cavity to radical procedures such as pericystectomy or hepatic resection . The type of surgery to be performed is determined by the location, size, and presence of cyst complications .

Cysto-biliary communication (CBC) is a common complication after hepatic HCD surgery that occurs when a cyst bursts into the biliary system , with a reported incidence of 13%-37% and can manifest as frank or occult (silent) CBC . Cyst fluid, scolices, small daughter cysts, and minor fragments of the endocyst membranes migrate into the biliary tract in occult or silent CBC, but neither clinically nor radiologically can be detected . Postoperative biliary leakage will occur if Occult CBC is overlooked during surgery, and will manifest as biliary drainage, biliary peritonitis, and biliary abscess. . Another issue is recurrence after hydatid cyst surgery, which has a range of (0-22 percent) .

Aim of the study, gap statement, and study strength:

Although several studies have looked at the results of laparoscopic partial cystectomy with omentoplasty in terms of postoperative biliary fistula and recurrence, no investigations into the link between occult cysto-biliary communication and late recurrence have been published. Furthermore, no studies have looked into the value of cystic fluid analysis in detecting occult cysto-biliary communication, which can lead to biliary leakage and recurrence after surgery. The primary goals of this study were to determine the prevalence and risk factors of occult CBC and recurrence, as well as the relationship between occult cysto-biliary communications manifested as postoperative biliary leakage and recurrence. The secondary goal was to use chemical analysis of hydatid cyst fluid to assess excessive bilirubin and alkaline phosphatase levels as predictors of fistula and recurrence.

Materials and methods:

Study design: This prospective multi-center experimental and follow-up study of six years duration was conducted at the hepato-biliary pancreatic units of our universities hospitals from September 2010 to September 2016. Initially, 292 patients were included, but only 244 patients enrolled in the final study as a comprehensive sample after the final assessment.

Participants: Stages CE2, CE3b According to the WHO-IWGE classification ,solitary, symptomatic or asymptomatic, superficial cyst, cases not suited for hepatic resection as the cyst wall abutting critical vascular and biliary structures as hepatic resection is harmful or excessive loss of hepatic tissue were used as inclusion criteria.The criteria for exclusion included the following: , stages CL, CE1, CE3a, CE4, CE5 according to WHO-IWGE classification of the hydatid cyst ,preoperative total bilirubin level greater than 2.0 mg/dl and direct bilirubin level greater than 1.5 mg/dl, common bile duct dilatation greater than 10 mm in the United States, or CT, or MRI, previous percutaneous treatment, recurrent cases after any type of surgery, cases with associated extrahepatic or extra-abdominal hydatid cyst, cysts affecting an entire lobe or the main pedicles, stages Cysts that are complicated (ruptured or diseased cysts), deep cysts, Patients who refuse intervention, have a surgical contraindication, are pregnant, have hydatid cysts in both lobes of the liver, previous liver surgery, liver abscess, frank CBC, cases lost during follow-up, cases who refused to take albendazole, or cases who developed albendazole-related issues (disturbed liver function).

Types of outcomes (study endpoints):

The primary outcomes were to determine the prevalence and risk factors of undetected cysto-biliary communication, recurrence, and the relationship between biliary fistula and recurrence. The secondary outcome was to see how well chemical analysis of hydatid cyst fluid might detect occult cysto-biliary problems and how they related to postoperative biliary leakage.

Definition of terms and measurement of outcomes:

An external biliary fistula Bile leakage was defined as a bilirubin concentration in the drain fluid of at least three times the serum bilirubin concentration on or after postoperative day three, or as the need for radiologic or operative intervention resulting from biliary collections or bile peritonitis, according to the International Study Group of Liver Surgery . The clinical care of patients with Grade A biliary leakage remains unchanged. Bile leakage in Grade B requires active therapeutic intervention but is treatable without relaparotomy, but bile leaking in Grade C necessitates relaparotomy.

Recurrence: is the appearance of new active cysts after intrahepatic or extrahepatic disease . Cysts areas imaged without a change in size and evidence of daughter cysts were not considered recurrence .

Postoperative morbidity: was evaluated by Clavien and Dindo . Hydatid cyst fluid analysis:Biochemical indexes of hydatid-cyst fluid detected by the automatic biochemical analyzer (AU-400, Olympus)

Recurrence-free survival is defined as the time from surgery until relapse of the disease at any site or death from any cause.

Perioperative technique and follow up:

All patients were assessed by multidisciplinary surgical, radiological, and anaesthetic teams prior to surgery. Liver function, serum alkaline phosphatase, and serum bilirubin were all tested before surgery, as well as the coagulation profile, ultrasound abdomen and pelvis, CT scan abdomen (Fig 1) and pelvis, and CT thorax. The protocol treatment for albendazole was 10mg/kg ten days prior to surgery and continued for six months after surgery with a two-week break between each month, with complete blood count and liver function tests. As in a prior study , a laparoscopic partial cystectomy with omentoplasty was performed.After the cystic cavity had been fully evacuated and complete hemostasis had been achieved, saline-soaked gauzes were placed in the cystic cavity for 10 minutes to observe the presence of bile while compressing either the gallbladder or common bile duct to stimulate bile backflow through cysto-biliary communication if present, and the visible orifices of the cystobiliary communications were oversewn. The process was completed if the gauzes were not stained with bile. A cholangiogram was not performed during the procedure.Omentoplasty was performed by inserting a right gastroepiploic-based flap from the larger omentum into the cavity and stitching it to the cyst wall with two to three interrupted vicryl 2/0 threads. In all cases, the subhepatic space was drained using a single drain. When there was no sign of bile leakage, a drain was routinely removed after 2-5 days. Patients were discharged home on the third and fifth postoperative days. Follow-up appointments were scheduled every one month, three months, six months, one year, and then every six months for the next four years, or if patients developed symptoms before the conclusion of the follow-up period (5 years). The bile drain was left open for a longer period of time in the case of bile drainage. Ultrasound was used to check the cyst cavity after surgery at 1, 3, 6 months, one year, and then every six months for the rest of the time. If the ultrasound results were inconclusive, a CT scan was ordered.

ELIGIBILITY:
Inclusion Criteria:

* Stages CE2
* CE3b According to the WHO-IWGE classification
* solitary
* symptomatic or asymptomatic
* superficial cyst
* cases not suited for hepatic resection as the cyst wall abutting critical vascular and biliary structures as hepatic resection is harmful or excessive loss of hepatic tissue

Exclusion Criteria:

* stages CL, CE1, CE3a, CE4, CE5 according to WHO-IWGE classification of the hydatid cyst
* preoperative total bilirubin level greater than 2.0 mg/dl and direct bilirubin level greater than 1.5 mg/dl
* common bile duct dilatation greater than 10 mm , or CT, or MRI, previous percutaneous treatment
* recurrent cases after any type of surgery, cases with associated extrahepatic or extra-abdominal hydatid cyst
* cysts affecting an entire lobe or the main pedicles
* stages Cysts that are complicated (ruptured or diseased cysts), deep cysts .Patients who refuse intervention, have a surgical contraindication, are pregnant, have hydatid cysts in both lobes of the liver, previous liver surgery, liver abscess, frank CBC, cases lost during follow-up, cases who refused to take albendazole, or cases who developed albendazole-related issues (disturbed liver function).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
biliary leakage | 30 days postoperatively
  incidence of biliary leakage detected clinically, sonar or CT
recurrence | 5 years
  detection of recurrence by CT and sonar abdomen

SECONDARY OUTCOMES:
biochemical analysis of hydatid cyst fluid | intraoperative
  estimation of bilirubin and alkaline phosphatase in cystic fluid by chemical analysis